CLINICAL TRIAL: NCT01019109
Title: Idiopathic Scoliosis Treated by Posterior Spinal Instrumentation. Evaluation of the 3D Correction, Aesthetic Outcomes and Quality of Life.
Brief Title: Scoliosis Surgery Using the PASS® LP System
Status: Completed | Type: Observational
Sponsor: Medicrea, USA Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: #0305
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Idiopathic Scoliosis
Keywords: scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Titanium rod: Titanium rods used as a part of PSF construct
  Interventions: Device: Posterior Spinal Fusion Device: Titanium rod arm used titanium rods, and CoCr rod arm used Cobalt Chrome rods as a part of the construct.
- CoCr Rod: Cobalt Chrome rods used as a part of PSF construct
  Interventions: Device: Posterior Spinal Fusion Device: Titanium rod arm used titanium rods, and CoCr rod arm used Cobalt Chrome rods as a part of the construct.

INTERVENTIONS:
Device: Posterior Spinal Fusion Device: Titanium rod arm used titanium rods, and CoCr rod arm used Cobalt Chrome rods as a part of the construct. — PASS LP Implant System is designed to contribute to correction and surgical stabilization of the thoracic, lumbar and sacral spine only. These implants are designed to stabilize the spine during normal development of solid bony consolidation which takes about 18 months. The internal fixation devices are composed of screws, hooks,rods, plates, cross links, connection and locking devices. The range of different sizes and shapes of the implants allows the surgeon to adapt to the pathology and morphology of each of his patients.
  Other Names: PASS® LP Spinal System; Low Profile Polyaxial Spine System; Pedicular Screw System

SUMMARY:
The purpose of this study is to find out the outcomes of using the PASS LP System to correct idiopathic scoliosis. This system is a unique set of spinal instrumentation used to surgically correct the rotation and deformity of the spine that is caused by scoliosis. Also, this study wants to find out the effects this system has on the physical appearance and quality of life for patients with scoliosis.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical, functional and radiographic outcomes following the reduction of idiopathic scoliosis.

The following will be evaluated

1. The 3D correction of scoliosis:

   * Reduction of scoliosis in the coronal plane (Cobb angles)
   * Correction in the sagittal plane (kyphotic and lordotic angles)
   * Correction of the axial vertebral rotation in the transverse plane
2. The functional and aesthetic outcomes

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic scoliosis requiring posterior spinal instrumentation and fusion
* Male and female

Exclusion criteria:

* Neuromuscular or degenerative scoliosis
* Spinal cord abnormalities with any neurologic symptoms or signs
* Spinal cord lesions requiring neurosurgical interventions, such as hydromyelia requiring Arnold Chiari decompression
* Primary muscle diseases, such as muscular dystrophy
* Neurologic diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, or spina bifida, Neurofibroma)
* Primary abnormalities of bones (e.g. osteogenesis imperfecta)
* Congenital scoliosis
* Scoliosis requiring anterior release
* Previous spinal surgery
* Patient who is unable to complete a self-administered patient questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgeon's Practice/Clinic
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Tridimensional radiographic correction of the scoliosis in coronal, sagittal and transverse planes | Preoperative, 6 weeks, 6 months, 1 year and 2 Years

SECONDARY OUTCOMES:
Functional and aesthetic outcomes | Preoperative, 6 months and 2 years
Perioperative and postoperative complications | Continuous during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Devito, M.D., Principal Investigator — Children's Healthcare of Atlanta, GA; Andrew King, M.D., Principal Investigator — LSU Health Sciences Center-New Orleans, LA; Mark Willits, M.D., Principal Investigator — Nationwide Children's Hospital- Columbus, OH; Afshin Aminian, MD, Principal Investigator — Chilren's Hospital of Orange County
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Nationwide Children's Hospital, Columbus, Ohio